CLINICAL TRIAL: NCT02531750
Title: Metabolic Complications Following Achilles Tendon Rupture - A Cohort Study
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kristoffer Barfod, MD, Hvidovre University Hospital
Other Study IDs: ATR_ORTHOMED
Record Dates: First submitted 2015-03-06; First posted 2015-08-24 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Achilles Tendon Rupture; Immobilization
Keywords: Metabolism; Bone metabolism; Glucose Metabolism; Lipid metabolism; Low grade inflamation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blod and urine samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Achilles tendon rupture: Patients with acute Achilles tendon rupture.
  Interventions: Other: Immobilization due to an Achilles tendon rupture

INTERVENTIONS:
Other: Immobilization due to an Achilles tendon rupture

SUMMARY:
Introduction This study will evaluate the effect on glucose, lipid and bone metabolism following conservative orthopaedic procedures in patients who suffered from acute Achilles tendon rupture. The sedentary rehabilitation period following these procedures may impact negatively upon glucose, lipid and bone metabolic pathways whereas the more physically active rehabilitation period instituted 8 weeks after the injury is hypothesized to impose positive metabolic effects.

The study is addition to the on-going clinical trial, Non-operative Treatment of Acute Achilles Tendon Rupture: Early Controlled Mobilization Compared With Immobilization, ClinicalTrials.gov Identifier: NCT02015364.

Perspective This study will establish whether the well-known effects on glucose, lipid and bone metabolism of a sedentary lifestyle can be observed already following 8 weeks of almost total abstain from physical activity in non-diabetic individuals, who suffered an acute Achilles tendon rupture. Thereby, we will add knowledge to the previous findings following strict bed-rest in healthy individuals on glucose and lipid metabolism and bone turnover. In a clinical perspective it is important to examine the extent to which individuals deteriorate in various metabolic pathways to better understand the pathophysiology behind these defects both in healthy individuals and in patients, who undergo bed rest or an equal reduction in physical activity as part of their rehabilitation.

Study design The present study includes 50 cases, who are examined early following injury (< 2 weeks) (baseline), 8 weeks (6 - 10 weeks) after injury and 52 weeks (40 - 64 weeks) after injury, respectively.

Oral glucose tolerance test (OGTT) with ingestion of 75 g of glucose during a maximum of 3 min from baseline (0 min). Plasma for glucose, insulin, C-peptide, NEFA will be drawn.

The individual will bring in morning spot urine for measurement of suPAR, creatinine, albumin and orosomucoid.

The individual will have drawn blood for measurement of HbA1c, total cholesterol, LDL cholesterol, HDL cholesterol, triglyceride, Na, K, creatinine, HgB, CRP, leukocytes, ALAT, alkaline phosphatase, Ca++, D vitamin, TSH, albumine and amylase. Also blood for BTM and plasma suPAR, IL6, TNFa and hsCRP will be drawn. Finally blood for lipid density profiling and lipid particle size will be drawn DXA of hip and lumbar spine including abdominal visceral and subcutaneous fat is done on a Hologic Discovery scanner.

DETAILED DESCRIPTION:
Introduction This study will evaluate the effect on glucose, lipid and bone metabolism following conservative orthopaedic procedures in patients who suffered from acute Achilles tendon rupture. The sedentary rehabilitation period following these procedures may impact negatively upon glucose, lipid and bone metabolic pathways whereas the more physically active rehabilitation period instituted 8 weeks after the injury is hypothesized to impose positive metabolic effects.

An on-going clinical trial, Non-operative Treatment of Acute Achilles Tendon Rupture: Early Controlled Mobilization Compared With Immobilization, ClinicalTrials.gov Identifier: NCT02015364 is already addressing as primary endpoints the Achilles tendon total rupture score and patient reported validation score developed to assess symptoms and physical activity after treatment for Achilles tendon rupture. The present study is an amendment/extension of that ongoing clinical trial.

An oral glucose tolerance test (OGTT) with frequent measurements of glucose, insulin, C-peptide and plasma free fatty acids can provide detailed information on insulin sensitivity, glucose tolerance, beta cell function, lipolysis and lipid oxidation as well as metabolic clearance of insulin(11-13).

Modern DXA scanners exhibit high performance and sensitivity to distinguish small changes in BMD. Also sensitive markers of changes in bone metabolism have recently been available. In particular two bone mass turnover markers (BTM) have been suggested to monitor bone resorption (CTX, carboxy-terminal cross-linked telopeptides of type 1 collagen) and bone formation ( P1NP, procollagen type 1 amino-terminal propeptide(14), but also osteocalcin (OC) is suggested as a marker of bone formation. DXA scanners have recently been validated to measure visceral adiposity, which is strongly associated with insulin sensitivity(15). A DXA scan exposes the individual to an X-ray radiation equal to only one day of background radiation, which makes this scanning modality much less harmful in terms of radiation dose compared to traditional CT scans (a 100-fold less radiation).

Traditional markers of low grade inflammation (LGI) include TNFa and IL6 and hsCRP. New promising markers include suPAR in plasma and urine and urine orosomucoid. suPAR has shown to predict CVD in non-diabetic community resting individuals(16). Urine orosomucoid is a strong predictor of major events in T2D and might be an early marker of glucose metabolic derangement(17). Low density lipoprotein (LDL) particles and especially those with a low particle size are atherogenic(18). Thus increased levels of LGI markers and immune markers including small LDL particles exhibit a particular at herogenic cocktail. A sedentary lifestyle is associated with an increase in these markers of LGI, impaired immune response and dyslipidaemia.

In the present setting we want to investigate the putative negative impact on glucose, lipid, and bone metabolism during a period of restrain from exercise secondary to immobilization following Achilles tendon rupture. We also want to study these patients during their physical active rehabilitation (at week 8 - 52), to establish whether they succeed in improving the metabolic impairments they suffered during the early post-injury period, during which period strong limitations in physical activity is prescribed (week 0 - 8).

Perspective This study will establish whether the well-known effects on glucose, lipid and bone metabolism of a sedentary lifestyle can be observed already following 8 weeks of almost total abstain from physical activity in non-diabetic individuals, who suffered an acute Achilles tendon rupture. Thereby, we will add knowledge to the previous findings following strict bed-rest in healthy individuals on glucose and lipid metabolism and bone turnover. In a clinical perspective it is important to examine the extent to which individuals deteriorate in various metabolic pathways to better understand the pathophysiology behind these defects both in healthy individuals and in patients, who undergo bed rest or an equal reduction in physical activity as part of their rehabilitation.

Hypothesis Implementation of a sedentary lifestyle with almost no physical activity in non-diabetic individuals undergoing non-operative treatment of acute Achilles tendon rupture will during 8 weeks

* impair insulin sensitivity and glucose effectiveness
* decrease disposition index
* compensatory decrease in insulin clearance
* decrease lipid oxidation
* increase visceral adipose tissue
* increase number of low density lipoprotein particles and a decrease the particle size
* increase immune and low grade inflammatory response as measured in plasma and urine
* induce bone loss in hip as measured by BMD
* increase bone resorption and decrease bone formation as measured by selected bone turnover markers.

During the following physical active rehabilitation from week 8 to week 52 the above proposed negative impact upon glucose, lipid and bone metabolism is thought to reverse at least partly so.

The relative positive effect on metabolic performance is hypothesized to be associated with duration from immobilization to full mobilization, which will be monitored by use of validated tools.

Study design Fifty non-diabetic individuals of age 18 to 70 years who should undergo non-operative treatment of acute Achilles tendon rupture and who are included to the randomized clinical trial: Non-operative Treatment of Acute Achilles Tendon Rupture: Early Controlled Mobilization Compared With Immobilization, ClinicalTrials.gov Identifier: NCT02015364 at the department of orthopaedics, Hvidovre Hospital are recruited as cases for this study. That study examines the effect on functional outcome measures of early controlled mobilization of the ankle from the beginning of week 3 following injury versus full immobilization during the initial 8 weeks post injury. Both groups are allowed full weight-bearing from the beginning of week 3 and physical activity level is expected to be the same in the two groups. As such randomization regime is unlikely to influence metabolism.

The present study includes 50 cases, who are examined early following injury (< 2 weeks) (baseline), 8 weeks (6 - 10 weeks) after injury and 52 weeks (40 - 64 weeks) after injury, respectively.

Examinations Oral glucose tolerance test (OGTT) with ingestion of 75 g of glucose during a maximum of 3 min from baseline (0 min). Plasma for glucose, insulin, C-peptide, NEFA will be drawn at time -10, -5, -1, 10, 15, 20, 30, 45, 60, 75, 90, 105, 120, 150, 180, 240 min. This test will be performed in the morning starting at approximately 8 am. The tests are done after an overnight fast of at least 10 hours.

The individual will bring in morning spot urine for measurement of suPAR, creatinine, albumin and orosomucoid.

Before the OGTT the individual will have drawn blood for measurement of HbA1c, total cholesterol, LDL cholesterol, HDL cholesterol, triglyceride, Na, K, creatinine, HgB, CRP, leukocytes, ALAT, alkaline phosphatase, Ca++, D vitamin, TSH, albumine and amylase. Also blood for BTM and plasma suPAR, IL6, TNFa and hsCRP will be drawn. Finally blood for lipid density profiling and lipid particle size will be drawn before the OGTT.

Body weight and height and waist and hip circumference will be measured. DXA of hip and lumbar columna including abdominal visceral and subcutaneous fat is done on a Hologic Discovery scanner by use of updated software. DXA will be carried out approximately at 12 am.

Acquisition of glucose and lipid metabolism will be done by use of the MinModel and the NEFA MinModel as described (11;12) All blood and urine samples will be destroyed after analysis. However a research biobank will be established since the period of time from most blood and urine sampling until analysis exceeds 1 week. This study will store all urine and blood samples in a freezer until all case subjects and controls have finished examinations. The duration of this period will be maximum 2 years from last patient last visit. Thus the research biobank will be established for storage only.

The urine and blood samples will be destroyed after analysis at Hvidovre and Glostrup Hospitals. Analysis results will all be anonymous and some will be sent abroad to our researcher Prof. Raymond Boston in USA, who will perform statistical calculations from analysis data. Permission for establishment of a research biobank is obtained from the Danish Data protection Agency.

Measurements of physical activity are acquired from the Primary Investigators ongoing trial "Non-operative Treatment of Acute Achilles Tendon Rupture: Early Controlled Mobilization Compared With Immobilization".

Statistics Ten days of bed rest in 13 healthy young individuals showed a 20% (P<0.05) significant decrease in insulin sensitivity and a 50% (P<0.05) reduction in lipid oxidation(2). Thirty-one days of bed rest in 8 healthy women was significantly associated with bone loss in total hip (2.07%, P<0.001)(7).

The present study does not imply strict bed rest but exhibits a longer sedentary period of following up compared to the above studies and include a larger number of participants, also. During the initial 8 weeks of strictly sedentary immobilization following the injury of the Achilles tendon we suggest that the patients will decrease their insulin sensitivity by at least 20%, the estimate of SD of the endpoint is 20%. Thus, using the MIREDIF statistics (Douglas Altman, Practical statistics for Medical research, Chapman & Hall, 1999), we can calculate that a population of 22 patients will generate a power >90% at significance level P<0.05 to investigate that primary endpoint. Similarly, the SD on lipidoxidation is 30% and the estimate is that the change during the sedentary period is at least 30%, thus by n=22 patients the power will be > 90%. Finally the change in BMD is likely 1% and the SD is 1%, thus n=22 patients will provide a statistical power of at least 90%. During the period of physical restitution we estimate a fully reversion of the deficit in endpoints during the sedentary period, i.e. similar calculation on power is valid during the restitution period.

The participants in the present study are included from the randomized clinical trial: Non-operative Treatment of Acute Achilles Tendon Rupture: Early Controlled Mobilization Compared with Immobilization. Randomization regime is unlikely to influence metabolism, however, it will be considered as a variable in the statistical analyses of the endpoints.

Ethical issues The study adheres to the Danish Act on Processing of Personal Data and, Danish Act on Health and the Helsinki II convention of clinical trials. All participants are informed about the purpose of the study and all ethical issues and a written consent is obtained before participation. At any given time, the participants can withdraw their acceptant for participation in the study. Personal data concerning demographic relations such as gender and age will be accessed as well to ensure the case subjects meet the inclusion criteria and for statistically use. To make assessments on study participation, the principal investigator will also gain access to relevant data from the patients medical files concerning illnesses or conditions the case subject might report.

The amount of blood drawn during the 52 weeks of participation in the study is less than 500 ml, which is the standard amount of blood drawn at a single donation of blood from a blood donor. The use of intravenous cannula can cause irritation or infection of vein or insertion site. All procedures will be performed as described in SOP.

The X-ray radiation from DXA during the study period equals 3 days of background radiation in Denmark and this amount of radiation is 30-fold less than that of a standard CT-scan of abdomen. In other words the dose of radiation is so low that a calculation of risk is not possible.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of age 18 to 70 years
* Rupture of Achilles tendon happened within 5 days.
* The patient must be expected to be able to attend rehabilitation and post-examinations.
* The patient must be able to speak and understand Danish.
* The patient must be able to give informed consent.

Exclusion Criteria:

* Former rupture of one or both Achilles tendon(s)
* Previous surgery on the Achilles tendon
* Fluoroquinolone treatment within the last 6 months
* Tendinosis treated with corticosteroids (tablets or injections) within the last 6 months.
* The patient has been diagnosed with arterial insufficiency in the legs.
* Terminal illness or severe medical illness: ASA score higher than or equal to 3.
* The space between the rupture and the calcaneus is less than 1cm.
* BMI >/= 35 kg/m2
* Known diabetes mellitus or HbA1c >/= 48 mol/mol
* Clinical significant anaemia, liver or kidney disease as judged by the sponsor or principal investigator.
* Thyroid function abnormality (TSH < 0.1 or TSH > 10)
* Calcium metabolic derangement, Ca++ < 1.1 or Ca++ > 1.40
* Known osteoporosis
* Re-rupture of the Achilles tendon between week 8 and 52

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty non-diabetic individuals of age 18 to 70 years who should undergo non-operative treatment of acute Achilles tendon rupture and who are included to the randomized clinical trial: Non-operative Treatment of Acute Achilles Tendon Rupture: Early Controlled Mobilization Compared With Immobilization, ClinicalTrials.gov Identifier: NCT02015364 at the department of orthopaedics, Hvidovre Hospital are recruited as cases for this study.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Glucose metabolism | Metabolic derangement: 0 to 8 weeks
  Insulin sensitivity as measured by MinModel-OGTT
Lipid metabolism | Metabolic derangement: 0 to 8 weeks
  Lipid oxidation as measured by MinModel-NEFA
Bone metabolism | Metabolic derangement: 0 to 8 weeks
  BMD changes in total hip
Atherosclerotic markers | Metabolic derangement: 0 to 8 weeks
  Changes in low density lipoprotein particles and in particle size

SECONDARY OUTCOMES:
Glucose metabolism | Metabolic derangement: 8 weeks; Metabolic restoration 52 weeks
  beta-cell responsiveness compared to insulin sensitivity (disposition index)
Glucose metabolism | Metabolic derangement: 8 weeks; Metabolic restoration 52 weeks
  glucose effectiveness
Glucose metabolism | Metabolic derangement: 8 weeks; Metabolic restoration 52 weeks
  insulin clearance
Glucose metabolism | Metabolic derangement: 8 weeks; Metabolic restoration 52 weeks
  changes in visceral adipose tissue
Lipid metabolism | Metabolic derangement: 8 weeks; Metabolic restoration 52 weeks
  changes in lipolysis
Lipid metabolism | Metabolic derangement: 8 weeks; Metabolic restoration 52 weeks
  changes in rates of which NEFA leaves plasma pool
Bone metabolism | Metabolic derangement: 8 weeks; Metabolic restoration 52 weeks
  changes in total BMD
Bone metabolism | Metabolic derangement: 8 weeks; Metabolic restoration 52 weeks
  changes in lumbar BMD
Bone metabolism | Metabolic derangement: 8 weeks; Metabolic restoration 52 weeks
  changes in BTM of bone resorption (CTX) and formation (P1NP, OC)
Atherosclerotic markers: Lipoproteins, immune response and low grade inflammation | Metabolic derangement: 8 weeks; Metabolic restoration 52 weeks
  changes in TNFa, IL6, hsCRP, suPAR and orosomucoid
Atherosclerotic markers: Lipoproteins, immune response and low grade inflammation | Metabolic derangement: 8 weeks; Metabolic restoration 52 weeks
  changes in density profiling of LDL and HDL cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer W Barfod, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Denmark